CLINICAL TRIAL: NCT04163874
Title: Alleviating Carbohydrate Counting for Patients With Type 1 Diabetes Using a Novel Insulin-plus-pramlintide Artificial Pancreas: a Randomized Controlled Crossover Trial.
Brief Title: Alleviating Carbohydrate Counting for Patients With Type 1 Diabetes Using a Novel Insulin-plus-pramlintide Artificial Pancreas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-5712
Record Dates: First submitted 2019-08-26; First posted 2019-11-15 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Type 1 Diabetes; Type 1 Diabetes Mellitus; Hyperglycemia, Postprandial
Keywords: type 1 diabetes; artificial pancreas; pramlintide; fiasp; hyperglycemia; closed-loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia | interventions — Insulin Aspart; pramlintide; Pancreas, Artificial

STUDY DESIGN:
Intervention Model Description: This is a three-way, randomized, blinded, crossover trial to compare the following strategies:
  (i) Fiasp-plus-Pramlintide closed-loop delivery with a simple meal announcement (pressing a button, no carbohydrate counting) (ii) Fiasp-plus-placebo closed-loop delivery with conventional carbohydrate counting (iii) Fiasp-plus-placebo closed-loop delivery with a simple meal announcement
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study will be a double-blinded study, where the participants and researchers will be blinded to the study drugs. Participants will wear two pumps for all interventions, one for insulin and the other for pramlintide/placebo (saline solution).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fiasp-plus-Placebo with Full Carbohydrate Counting (Experimental): Fiasp insulin and placebo insulin infusion in two insulin pumps with full carbohydrate counting.
  Interventions: Drug: Fiasp; Drug: Placebo; Device: Artificial Pancreas
- Fiasp-plus-placebo with Simple Meal Announcement (Placebo Comparator): Fiasp insulin and placebo (saline) insulin infusion in two insulin pumps using the simple meal announcement system.
  Interventions: Drug: Fiasp; Drug: Placebo; Device: Artificial Pancreas
- Fiasp-plus-Pramlintide with Simple Meal Announcement (Active Comparator): Fiasp insulin and pramlintide insulin infusion in two insulin pumps using the simple meal announcement system.
  Interventions: Drug: Fiasp; Drug: Pramlintide Acetate; Device: Artificial Pancreas

INTERVENTIONS:
Drug: Fiasp — Fiasp Insulin delivered in a basal-bolus manner.
Drug: Pramlintide Acetate — Pramlintide delivered in a basal-bolus manner with a fixed ratio with insulin.
  Arms: Fiasp-plus-Pramlintide with Simple Meal Announcement
Drug: Placebo — Placebo delivered in a basal-bolus manner with a fixed ratio with insulin.
  Arms: Fiasp-plus-Placebo with Full Carbohydrate Counting; Fiasp-plus-placebo with Simple Meal Announcement
Device: Artificial Pancreas — Tandem insulin pump, dexcom G5 sensor, Nexus 5 cellphone running the iMAP algorithm.

SUMMARY:
One of the main challenges in maintaining tight glucose control in a closed-loop system occurs at meal times. Amylin is a gluco-regulatory beta-cell hormone that is co-secreted with insulin in response to nutrient stimuli, and is deficient in patients with type 1 diabetes. Amylin, in the postprandial period, contributes to regulating glucose levels by delaying gastric emptying, suppressing nutrient-stimulated glucagon secretion, and increasing satiety. Pramlintide is a synthetic analog of the hormone amylin. A closed-loop system that delivers both insulin and pramlintide, based on glucose sensor readings, has the potential to better normalize glucose levels, especially during the post-prandial period.

The aim of this project is to assess whether co-administration of pramlintide with the improved insulin aspart formulation - Fiasp, in an artificial pancreas system, will alleviate the need for carb counting by replacing it with a simple meal announcement, without degrading the quality of glycemic control in a closed-loop therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent
2. Males and females ≥ 12 years of age
3. HbA1c ≤ 12%
4. Insulin pump use for at least 3 months
5. Clinical diagnosis with type 1 diabetes for at least 12 months. The diagnosis of T1D is based on the investigator's clinical judgment; C peptide level and antibody determinations are not planned.
6. Women of child-bearing potential must be ready and able to use a highly effective method of birth control. Women of childbearing potential are females who have experienced [the first occurrence of menstruation] and do not meet the criteria for women not of childbearing potential. Women not of childbearing potential are females who are permanently sterile or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause.

Exclusion Criteria:

Participants who meet any of the following criteria are not eligible for the study:

1. Current or ≤ 1 month use of other antihyperglycemic agents (SGLT2 inhibitors, GLP-1 agonists, Metformin, Acarbose, etc.…).
2. Current use of glucocorticoid medication.
3. Use of medication that alters gastrointestinal motility.
4. Planned or ongoing pregnancy.
5. Breastfeeding individuals.
6. Severe hypoglycemic episode within one month of admission.
7. Severe diabetes ketoacidosis episode within one month of admission.
8. Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
9. Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
10. Known hypersensitivity to any of the study drugs or their excipients.
11. Individuals with confirmed gastroparesis.
12. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
13. Unable to travel to research center within 3h if needed during study interventions
14. Failure to comply with team's recommendations (e.g. not willing to eat meals/snacks, not willing to change pump parameters, etc.).

Study Discontinuation/Withdrawal

1. Failure to comply with the protocol.
2. Pregnancy.
3. After an event which the PI believes it is not in the best interest for the patient to continue the trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Each participant's time in target range | 12 days
  Time in target range (3.9-10mmol/L)
Mean score of the Emotional Burden section of the Diabetes Distress Scale | 12 days
  Average of all question's scores (from 1-6). Higher score means more emotional burden.

SECONDARY OUTCOMES:
Each participant's percentage of time of glucose levels spent between 3.9 and 7.8 mmol/L | 12 days
Each participant's percentage of time of glucose levels spent between 3.9 and 10 mmol/L | 12 days
Each participant's percentage of time of glucose levels spent below 3.9, 3.3, and 2.8 mmol/L | 12 days
Each participant's percentage of time of glucose levels spent above 7.8, 10, 13.9 and 16.7 mmol/L | 12 days
Each participant's mean glucose level | 12 days
Each participant's standard deviation of glucose levels as a measure of glucose variability | 12 days
Each participant's number of hypoglycemia events defined as at least 15 min below 3.0 mmol/L | 12 days
Each participant's number of Gastrointestinal symptoms | 12 days
Each participant's total insulin delivery | 12 days

CONTACTS AND LOCATIONS:
Locations (1):
- 3555 University Street, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The raw data (i.e., insulin delivery, glucose levels, individual participant data) and informed consent form could be shared by the corresponding author, ahmad.haidar@mcgill.ca, upon reasonable request for academic purposes, subject to Material Transfer Agreement and approval of McGill University Health Center's Research Ethics Board. All data shared will be deidentified. Study protocol is available with publication.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Cohen E, Tsoukas MA, Legault L, Vallis M, Von Oettingen JE, Palisaitis E, Odabassian M, Yale JF, Garfield N, Gouchie-Provencher N, Rutkowski J, Jafar A, Ghanbari M, Haidar A. Simple meal announcements and pramlintide delivery versus carbohydrate counting in type 1 diabetes with automated fast-acting insulin aspart delivery: a randomised crossover trial in Montreal, Canada. Lancet Digit Health. 2024 Jul;6(7):e489-e499. doi: 10.1016/S2589-7500(24)00092-X. PMID 38906614